CLINICAL TRIAL: NCT07091539
Title: Food Insecurity and MASLD: A Fruit and Vegetable Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Gastroenterological Association (Other); University of California, San Francisco Population Health Health Equity Award (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-42019
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Food Insecurity Among Children
Keywords: MASLD; Food insecurity; pediatrics
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with MASLD and food insecurity (Experimental): This group will receive $80 of fruit/vegetable vouchers per month x 6 months; parents/ guardians will participate in a semi-structured interview at the end of the study
  Interventions: Other: Fruit/vegetable vouchers

INTERVENTIONS:
Other: Fruit/vegetable vouchers — The intervention is $80 of fruit/vegetable vouchers (EatSF Veggies4Vouchers) per month x 6 months

SUMMARY:
This proposal addresses a critical gap in the understanding of the impact of household food insecurity (FI) on pediatric metabolic dysfunction-associated steatotic liver disease (MASLD) severity. Evidence from adult studies links household FI to MASLD and liver fibrosis, and prior research of the PI has shown that exposure to household FI in early childhood was associated with a nearly fourfold increased odds of pediatric MASLD in middle childhood. Possible mechanisms linking household FI to pediatric MASLD include lower intake of fruits and vegetables, higher intake of caloric dense nutrient-poor foods (e.g., sugar-sweetened beverages), and less diversity of foods. Given consensus recommendations for the management of MASLD focus on lifestyle modification, i.e., diet and exercise to achieve weight loss, this proposal seeks to assess whether a clinic-based fruit/vegetable voucher intervention program (EatSF) could potentially improve clinical outcomes for children/adolescents with MASLD and household FI. Study participants include children/adolescents with household FI and MASLD who are receiving care at UCSF's liver clinic and Weight Management for Teen and Child Health (WATCH) Clinic, a pediatric subspecialty clinic. The study seeks to identify barriers and facilitators to fruit/vegetable voucher redemption, and assess changes in dietary intake, MASLD severity, and other cardiometabolic health factors in children participating in the pilot intervention. Study findings will form the basis of an R01 application to conduct a fully powered randomized controlled trial of the intervention.

DETAILED DESCRIPTION:
Study designs for each of the three specific aims are below:

Aim 1: Assess participation in the EatSF intervention (to be piloted in the liver and WATCH clinics) among families with a child with MASLD and household FI, as identified through an observational cross-sectional study.

Design: To achieve this aim, the investigators will conduct a 6-month pre-post one-arm pilot intervention study of the EatSF Vouchers4Veggies fruit and voucher program with families with a child with household FI and MASLD who receive care at the UCSF liver or WATCH Clinics. At the end of the 6-month intervention period, the investigators will assess the percentage of vouchers redeemed through a software program developed by EatSF Vouchers4Veggies. Also at the end of the 6-month intervention, the CRC will administer study assessments comparable to those conducted at baseline as part of the observational cross-sectional study (for which IRB approval has been submitted). Also at the end of the 6-month intervention, the CRC will conduct semi-structured interviews to identify barriers and facilitators to:

1. voucher redemption,
2. adhering to clinic dietary recommendations, and
3. parental understanding of MASLD and the role of diet in its management.

Aim 2: Assess changes in dietary intake in children with MASLD and FI participating in the 6-month pre-post one-arm pilot intervention study with families with a child with household FI and MASLD who receive care at the UCSF liver or WATCH Clinics (projected n=48).

Design: To achieve this aim, the investigators will analyze changes in the baseline data collected as part of the observational cross-sectional study (for which IRB approval has been submitted) with post-test data (collected at the end of the six-month pilot study).

Exploratory Aim 3: Assess changes in liver inflammation measured by alanine aminotransferase serum lab (ALT) (GGT), and other cardiometabolic health factors in children with MASLD and household FI from baseline to the end of the 6-month study.

Design: To achieve this aim, the investigators will analyze data collected from the 6-month pre-post one-arm pilot intervention study with families with a child with household FI and MASLD who receive care at UCSF's liver and WATCH clinics.

ELIGIBILITY:
Inclusion Criteria:

* The study population for all study aims consists of children and adolescents receiving care at the liver and WATCH clinics.

Inclusion criteria include:

* family living in California;
* a parent/guardian who speaks Spanish or English,
* child is between the ages of 6 to <18 years;
* child has elevated BMI greater than or equal to 85% for age and sex
* child has ALT value greater than 26 for boys and 22 for girls on two occasions within the last year; OR one elevated ALT value and imaging confirming steatosis
* family does not intend to move out of California for the next year;
* family is not already receiving EatSF Fruit and Vegetable Vouchers;
* family is not participating in any other dietary education programs besides that offered by the liver/ WATCH clinics

Exclusion Criteria:

* child has an underlying condition or medication causing their weight gain (i.e., hypothyroidism, Prader-Willi syndrome, antipsychotic medications) or a known liver condition other than MASLD/MASH causing their elevated liver numbers;
* child is on a weight loss medication (including: Qsymia or GLP-1 receptor agonists),
* both of which are assessed as part of routine clinical care.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Voucher participation | From enrollment to the end of the six month intervention
  What percentage of money of the vouchers were used monthly
Changes in dietary intake | From baseline to the end of the six month intervention
  Assess changes in dietary intake in children with MASLD and FI participating in the 6 month pre-post one arm pilot intervention studies.
changes in liver inflammation and other cardiometabolic health factors | From baseline to the end of the six months study.
  Assess changes in liver inflammation as measured by ALT and GGT and other cardiometabolic health factors in children with MASLD and FI from baseline to the end of the six months study.

OTHER OUTCOMES:
Semi-structured interviews | At the end of the six month intervention
  At the end of the six months, semi-structured interviews will be conducted to identify barriers and facilitators to voucher redemption, adhering to clinic recommendations, and to explore the parental understanding of MASLD and the role of diet in its management.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Maxwell, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maxwell SL, Price JC, Perito ER, Rosenthal P, Wojcicki JM. Food insecurity is a risk factor for metabolic dysfunction-associated steatotic liver disease in Latinx children. Pediatr Obes. 2024 Jun;19(6):e13109. doi: 10.1111/ijpo.13109. Epub 2024 Mar 7. PMID 38453472
- [Background] Landry MJ, van den Berg AE, Asigbee FM, Vandyousefi S, Ghaddar R, Davis JN. Child-Report of Food Insecurity Is Associated with Diet Quality in Children. Nutrients. 2019 Jul 12;11(7):1574. doi: 10.3390/nu11071574. PMID 31336880
- [Background] Kardashian A, Dodge JL, Terrault NA. Racial and ethnic differences in diet quality and food insecurity among adults with fatty liver and significant fibrosis: a U.S. population-based study. Aliment Pharmacol Ther. 2022 Nov;56(9):1383-1393. doi: 10.1111/apt.17219. Epub 2022 Sep 29. PMID 36173037
- [Background] Kardashian A, Dodge JL, Terrault NA. Food Insecurity is Associated With Mortality Among U.S. Adults With Nonalcoholic Fatty Liver Disease and Advanced Fibrosis. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2790-2799.e4. doi: 10.1016/j.cgh.2021.11.029. Epub 2021 Dec 16. PMID 34958747
- [Background] Tamargo JA, Sherman KE, Campa A, Martinez SS, Li T, Hernandez J, Teeman C, Mandler RN, Chen J, Ehman RL, Baum MK. Food insecurity is associated with magnetic resonance-determined nonalcoholic fatty liver and liver fibrosis in low-income, middle-aged adults with and without HIV. Am J Clin Nutr. 2021 Mar 11;113(3):593-601. doi: 10.1093/ajcn/nqaa362. PMID 33515016
- [Background] Golovaty I, Tien PC, Price JC, Sheira L, Seligman H, Weiser SD. Food Insecurity May Be an Independent Risk Factor Associated with Nonalcoholic Fatty Liver Disease among Low-Income Adults in the United States. J Nutr. 2020 Jan 1;150(1):91-98. doi: 10.1093/jn/nxz212. PMID 31504710